CLINICAL TRIAL: NCT06517381
Title: Awareness About Warning Signs of Mental Illness Using Social Media Among Health Professions' Students in Saudi Arabia: A Quasi Experimental Study
Brief Title: Awareness About Warning Signs of Mental Illness Among Health Profession Students. A Quasi-Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud Bin Abdulaziz University for Health Sciences (Other)
Responsible Party: Principal Investigator, Abeer Selim, Assistant Professor, King Saud Bin Abdulaziz University for Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-01-R-005
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Online Warning Signs of Mental Illness Literacy Program (Experimental): 30-minute pre-recorded educational video with interactive question-and-answer sessions
  Interventions: Other: Digital Online Warning Signs of Mental Illness Literacy Program

INTERVENTIONS:
Other: Digital Online Warning Signs of Mental Illness Literacy Program — Digital Online Warning Signs of Mental Illness Literacy Program is comprised of 30-minute pre-recorded video and question-and-answer sessions. The videos were followed by case studies, success stories, and interactive question-and-answer sessions

SUMMARY:
In Saudi Arabia, there are limited studies addressing mental health literacy, with no studies regarding warning signs of mental illness. Mental health literacy among healthcare professions students as future clinicians decreases stigma and promotes mental health through early detection and management of mental health problems.

The current study aimed to evaluate the effectiveness of a digital online educational session about the warning signs of mental illness called the Digital Base Warning Signs of Mental Illness Literacy Program.

This study hypothesized that the Digital Base Warning Signs of Mental Illness Literacy Program is effective and will enhance health profession students' literacy regarding warning signs of mental illness.

This is a non-randomized trial using a 30-minute digital educational session about the warning signs of mental illness. It involves a convenience sample of 493 undergraduate health profession students. The Mental Health Literacy Survey About Warning Signs of Mental Illness was developed and validated to measure the participants' mental health literacy before and after the intervention.

DETAILED DESCRIPTION:
Improving warning signs of mental health literacy is a critical focus for this study as it addresses the fundamental understanding and recognition of early indicators of mental health issues. This first-of-its-kind study aims to fill a significant gap in current research by systematically examining the effectiveness of targeted interventions designed to enhance awareness and comprehension of mental health warning signs. Effective management of mental health issues among university students requires early detection of warning signs of mental illnesses and access to treatment to improve individuals' psychological, academic, social, and occupational functioning.

The current study aimed to evaluate the effectiveness of a digital online educational session about the warning signs of mental illness called the Digital Base Warning Signs of Mental Illness Literacy Program.

This study hypothesized that the Digital Base Warning Signs of Mental Illness Literacy Program is effective and will enhance health profession students' literacy regarding warning signs of mental illness.

The current study used a quasi-experimental nonrandomized trial, one-group pretest-posttest study design, which used Transparent Reporting of Evaluation with Nonrandomised Designs.

TOOLS Sociodemographic questions Items included age, gender, college, academic year, type of university, knowing anyone who has mental illness, and experience of mental illness.

Mental Health Literacy Survey About Warning Signs of Mental Illness After reviewing the literature, the researchers developed the survey to measure participants' mental health literacy about the warning signs of mental illness. The tool was created because the existing instruments do not adequately capture the specific contents and indicators pertinent to mental health literacy about warning signs of mental illness. Moreover, having a standardized tool allows for consistent data collection and comparison across different populations and settings, which is vital for advancing mental health literacy research and enabling researchers to draw more accurate conclusions and develop evidence-based recommendations.

The survey has 15 items, each measuring agreement on a five-point Likert scale, ranging from strongly agree to strongly disagree). The survey scores ranged from 15 (Lowest) to 75 (Highest). Items from 1 to 11 address knowledge about warning signs of mental illness, tackling social withdrawal, impairment in academic or occupational functioning, cognitive impairment, perceptual hypersensitivity, avolition or apathy, dissociation or sense of unreality, unusual beliefs, suspiciousness, odd behaviors, marked changes in sleep or appetite or deterioration of hygiene, and mood swings. Items from 12 to 15 are related to early detection, utilization of mental health resources, and attitudes toward mental illness. The Survey underwent a validation process. After developing MHLS, content validity was established, and after data collection, construct validity was measured using factor analysis.

INTERVENTION Digital Online Warning Signs of Mental Illness Literacy Program The investigators developed the program in collaboration with the university media center. The program comprised 30-minute pre-recorded video and question-and-answer sessions. Previous studies have demonstrated the effectiveness of educational programs lasting between 30 and 45 minutes in enhancing nurses' knowledge and practices. The video sessions demonstrated motion graphic animation of 11 warning signs of mental illness: social withdrawal, impairment in academic or occupational functioning, cognitive impairment, perceptual hypersensitivity, avolition or apathy, dissociation or sense of unreality, unusual beliefs, suspiciousness, odd behaviors, marked changes in sleep or appetite or deterioration of hygiene, and mood swings. After demonstrating warning signs of mental illness, the video showed that experiencing several of the earlier symptoms that seriously impair social, academic, or occupational functioning needs mental health consultation. Further, the video emphasized that untreated warning signs might develop into psychotic episodes. After that, pharmacological and nonpharmacological therapies were presented. Furthermore, the significance of early intervention in managing mental illness and preventing further disabilities, as in the case of physical disorders, was illustrated. The videos were followed by case studies, success stories, and interactive question-and-answer sessions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female university health professional students

Exclusion Criteria:

* Other university specialty students

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 494 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Recognizing Warning Signs of Mental Illness | Once the intervention is completed/immediately after the intervention
  students will be able to identify warning signs of mental illness and understand the significance of early recognition measured byMental Health Literacy Survey About Warning Signs of Mental Illness scoring ranges from 15 to 75

CONTACTS AND LOCATIONS:
Overall Officials: ABEER SELIM, RN, PhD, Principal Investigator — College of Nursing-Riyadh, King Saud Bin Abdulaziz University for Health Sciences
Locations (2):
- Saudi Arabia (2):
  - King Abdullah International Medical Research Center, Riyadh
  - King Saud bin Abdulaziz University for health sciences, Riyadh

IPD SHARING:
Plan to Share IPD: Yes
Unidentified data will shared with other researchers contributing to this study to analyze data, present results, and interpret the results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2022 - July 2024
Access Criteria: Study investigators